CLINICAL TRIAL: NCT06208696
Title: Pilot Study to Evaluate the Role of an Evidenced-based Chronic-disease Self-management Program to Support Challenges Experiencing Patients Living With Long-COVID and Chronic Diseases in Puerto Rico
Brief Title: Chronic-disease Self-management Program in Patients Living With Long-COVID in Puerto Rico
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Puerto Rico (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Enid J. Garcia-Rivera, Associate Professor, University of Puerto Rico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2309143222; SubOTA 6922-03-COVID-S026 (Other Grant/Funding Number: UPRCCC)
Record Dates: First submitted 2023-12-11; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Long Covid19
Keywords: Long COVID19; chronic disease self-management; evidenced-based program; health-related quality of life
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: The intervention group will participate in an evidenced-based intervention from chronic disease self-management and the control group will receive usual care and published information for chronic disease management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (TCS) (Experimental): Participants with Long-COVID and chronic diseases that agree to participate in the intervention will participate in the "Tomando Control de su Salud" (TCS) workshops. TCS is an evidenced based intervention in Spanish and a culturally appropriate version similar to the Chronic Disease Self-Management program of the Centers for Disease Control and Prevention (CDC) aimed to improve disease management skills, including decision making, problem solving, and action planning among patients with at least one chronic condition.
  Interventions: Other: "Tomando control de su salud" (Spanish Chronic Disease Self-Management)
- Non-Intervention Group (Regular care) (No Intervention): Those not interested in participating in the intervention will receive general information about chronic disease management available at the CDC website in Spanish, by email or in person.

INTERVENTIONS:
Other: "Tomando control de su salud" (Spanish Chronic Disease Self-Management) — "Tomando control de su salud" (Spanish Chronic Disease Self-Management) is a culturally appropriate program developed in Spanish to support Hispanics patients to build confidence in their ability to manage their health. This intervention was developed by Lorig et al. at Stanford University and has been widely used by the Puerto Rico Department of Health since it is recommended by the CDC as an evidenced-based intervention for chronic disease management.
  Arms: Intervention group (TCS)

SUMMARY:
This is a pilot non-randomized-controlled trial to evaluate the impact of "Tomando control de su salud", an evidenced-based intervention for chronic disease self-management in the quality of life of patients living with Long-COVID in Puerto Rico.

DETAILED DESCRIPTION:
Patients from our cohort study entitle "The Puerto Rico COVID-19 Assessment Study" (PR-COAS) (IRB# 2290030465) will be invited to participate in this pilot study during the 12-month follow-up call. Participants with long-COVID and at least one chronic diseases that agree to participate in the pilot study will be allocated into one of the study intervention groups that will participate in the "Tomando Control de su Salud" (TCS) workshops. This group will be asked to answer a final interview approximately one month after the last workshop. Those not interested in participating in the intervention will receive general information about chronic disease management available at the CDC website in Spanish, by email or in person, in addition to their regular health care and will be asked to answer the interview approximately 3 months after the last interview of the PR COAS-cohort.

Investigators expect to enroll approximately 50 participants that will be divide between the groups of intervention and non-intervention. Participants will receive an incentive for transportation and/or parking expenses and for the time dedicated for their participation.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 21 years or older;
2. Participant of PR COAS-cohort that completed the last interview (12-month-follow-up) and authorized to be contacted for further studies;
3. Having at least one chronic condition (excluding cancer) diagnosed by a physician or healthcare provider, and
4. Ability to attend weekly sessions.

Exclusion Criteria:

1. Any clinical or cognitive impairment that limits the participant's ability to decide to participate in the study or complete the interviews;
2. presence of a life threatening or extreme medical condition, and
3. planning to move out of the municipality within the next year.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of the impact of health-related quality of life | 1-3 months
  The following EuroQol (EQ) instrument is used: EQ-5D-5L (Spanish version) scale. This instrument measures quality of life on five dimensions: mobility, self-care, daily activities, pain or discomfort, and anxiety or depression. Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5).
Assessment of the fatigue in the impact of the health-related quality of life | 1-3 months
  The investigators use the Fatigue questionnaire (NIH PROMIS© Neuro-QoL Item Bank v1.0, Short Form, Spanish version).
Assessment of the Post-COVID 19 in the impact of health-related quality of life | 1-3 months
  Investigators uses the Post-COVID-19 Functional Status Scale (PCFS, Spanish version). An ordinal tool that focuses on relevant aspects of daily life during follow-up after the COVID-19 infection (Klok et al., 2020). PCFS includes the entire range of functional outcomes by focusing on limitations (if any) in usual duties/activities either at home or at work/study, as well as changes in lifestyle.
Assessment of the anxiety in the impact of health-related quality of life | 1-3 months
  Anxiety (GAD-7, Spanish version) - It is a validated one-dimensional 7-item questionnaire for generalized anxiety disorder assessment, as listed in the DSM-IV.

SECONDARY OUTCOMES:
Chronic diseases self-management | 1-3 months
  Chronic diseases self-management will be assessed through the following scales:
  Self-Care of Chronic Illness Inventory (SC-CII v4.c, Spanish version): It is an internationally generic measure used to assess self-care in chronic diseases, and it is based on the Theory of Self-Care of Chronic Illness. SC-CII comprises four scales: self-care maintenance (Section A), self-care monitoring (Section B), self-care management (Section C), and self-care confidence (Section D) 31. For the study, investigators will just use the first three sections of this instrument.
Auto-efficacy for disease management | 1-3 months
  Auto-efficacy will be assessed through the following scales:
  NIH PROMIS© 4-item Short Forms v1.0, 4a - Self-Efficacy for Managing Chronic Conditions, which is a multidimensional categorical model to estimate individual's self-efficacy for managing their heath chronic diseases through the following five behavioral domains:Self-Efficacy for Managing Daily Activities, Self-Efficacy for Managing Emotions, Self-Efficacy for Managing Medications and Treatments, Self-Efficacy for Managing Social Interactions, Self-Efficacy for Managing Symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Enid J Garcia-Rivera, MD, MPH, Principal Investigator — University of Puerto Rico Medical Sciences Campus
Locations (1):
- Centro Dotal de Investigaciones de Servicios de Salud, UPR-MSC (Hospital UPR), Carolina, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu DS, De Maria M, Barbaranelli C, Vellone E, Matarese M, Ausili D, Rejane RE, Osokpo OH, Riegel B. Cross-cultural applicability of the Self-Care Self-Efficacy Scale in a multi-national study. J Adv Nurs. 2021 Feb;77(2):681-692. doi: 10.1111/jan.14617. Epub 2020 Dec 9. PMID 33295675
- [Background] Lorig KR, Ritter PL, Gonzalez VM. Hispanic chronic disease self-management: a randomized community-based outcome trial. Nurs Res. 2003 Nov-Dec;52(6):361-9. doi: 10.1097/00006199-200311000-00003. PMID 14639082
- See also: Johns Hopkins University, Center for Systems Science and Engineering COVID19 Dashboard. — https://coronavirus.jhu.edu/map.html
- See also: Dong, E., Du, H., & Gardner, L. (2020). An interactive web-based dashboard to track COVID-19 in real time. The Lancet infectious diseases, 20(5), 533-534. — https://doi.org/10.1016/S1473-3099(20)30120-1
- See also: Soriano, J. B., Murthy, S., Marshall, J. C., Relan, P., & Diaz, J. V. (2022). A clinical case definition of post-COVID-19 condition by a Delphi consensus. The Lancet Infectious Diseases, 22(4), e102-e107. ISSN 1473-3099. — https://doi.org/10.1016/S1473-3099(21)00703-9
- See also: Davis, H. E., Assaf, G. S., McCorkell, L., Wei, H., Low, R. J., Re'em, Y., ... & Akrami, A. (2021). Characterizing long COVID in an international cohort: 7 months of symptoms and their impact. EClinicalMedicine, 38, 101019, ISSN 2589-5370. — https://doi.org/10.1016/j.eclinm.2021.101019
- See also: Physical and mental health 3 months after SARS-CoV-2 infection (long COVID) among adolescents in England (CLoCk): A national matched cohort study, The Lancet Child & Adolescent Health, 6(4), 230-239. — https://doi.org/10.1016/S2352-4642(22)00022-0
- See also: Yang, C., Zhao, H., & Tebbutt, S. J. (2021). Long-term effects on survivors with COVID-19. The Lancet, 398(10314), 1872. — https://doi.org/10.1016/S0140-6736(21)02323-0
- See also: National Institutes of Health. (2021). RECOVER: A Multi-site Observational Study of Post-Acute Sequelae of SARS-CoV-2 Infection in Adults Version 3.0. Accessed 6 April 2022. — https://recovercovid.org
- See also: US Department of Health and Human Services. National Institutes of Health (2022). Patient-reported Outcomes Measure Information Systems (PROMIS). — https://commonfund.nih.gov/promis/index
- See also: EuroQolResearchFoundation (2019). EQ-5D-5L User Guide: Basic information on how to use the EQ-5D-5L instrument, version 3.0. — https://euroqol.org/publications/user-guides
- See also: Riegel, B. (Author) & Jose, M. M. (Translator). (nd). Self-Care Self-Efficacy Scale (Spanish). — https://self-care-measures.com/project/self-care-self-efficacy-scale-spanish-2/
- See also: U. S. Department of Health and Human Services. (2017). PROMIS® (Patient-Reported Outcomes Measurement Information System) Health Measures: Self-Efficacy for Managing Chronic Conditions. PROMIS Item Bank v1.0, Short Forms 4a. — https://www.healthmeasures.net/indexphp?option=com_instruments&task=Search.pagination&Itemid=992
- See also: Johns Hopkins Bloomberg School of Public Health. (nd). COVID-19 Community Response Survey. Module 5 Comorbidities and Care Engagement. Protocol - Health Conditions, Medications and Health Care during COVID-19 Pandemic (PhenX Toolkit). — https://www.phenxtoolkit.org/protocols/view/940301?origin=subcollection
- See also: Johns Hopkins Bloomberg School of Public Health. (2020). COVID-19 Research: History, Treatment and Outcomes. Protocol - Access to Health Services (Spanish version), CDC National Health Interview Survey (NHIS) Utilization Questionnaire, 2020. — https://www.phenxtoolkit.org/protocols/view/270101?origin=subcollection
- See also: US Centers for Disease Control and Prevention (2021). Cuestionario del BRFSS 2020. — https://www.cdc.gov/brfss/questionnaires/pdf-ques/2020-brfss-questionnaire-spanish-verison-508.pdf
- See also: GAD-7 (Spanish version). — https://didihirsch.org/wp-content/uploads/GAD-7-Generalized-Anxiety-Disorder-Spanish.pdf